CLINICAL TRIAL: NCT05218304
Title: Baromètre Santé Adulte 2021-2022 in People Aged 18 to 64 in New Caledonia Using the WHO STEPwise Approach
Brief Title: Baromètre Santé Adulte 2021-2022
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lockdown in the general population due to COVID
Sponsor: Agence Sanitaire et Sociale de Nouvelle Calédonie (Other Government)
Collaborators: Institut Pasteur (Industry); Pacific Community (Other); World Health Organization (Other); Institut de la Statitique et des Etudes Economiques Nouvelle Calédonie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2021-A01260-41
Record Dates: First submitted 2022-01-18; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Diabetes; Hypercholesterolemia; Renal Failure; Dengue Fever; Zika; Chikungunya; Ross River; Malaria; SARS-CoV Infection; Chronic Disease
Keywords: Chronic disease; Diabetes; WHO STEP approach; Prevalence; New Caledonia
MeSH Terms: conditions — Diabetes Mellitus; Hypercholesterolemia; Renal Insufficiency; Dengue; Zika Virus Infection; Chikungunya Fever; Ross River Virus Infection; Malaria; Severe Acute Respiratory Syndrome; Chronic Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is an observational, descriptive and cross-sectional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sample (No Intervention): questionnaires physical measurements (height, weight, perimeter abdominal and blood pressure)
- Sub-sample - blood test (Experimental): questionnaires physical measurements (height, weight, perimeter abdominal and blood pressure) Blood samples
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — A questionnaire, physical measurements (height, weight, perimeter abdominal and blood pressure) for all arm will be done, approximately 5400 people carried out by investigators. Only 1800 will undergo blood samples carried out by nurses
  Arms: Sub-sample - blood test

SUMMARY:
In 2021-2022, Agence Sanitaire et Sociale Nouvelle Calédonie (ASSNC) is undertaking the "Baromètre Santé Adulte" for the third time. This study is carried out this year in collaboration with WHO and Institut Pasteur de Nouvelle Calédonie (IPNC).

The main objective of this investigation is to describe the current levels of chronic disease risk factors in the adult population of New Caledonia aged from 18 to 64 years old. This study will also help to estimate prevalence of certain diseases (diabetes, hypercholesterolemia, renal failure), seroprevalence of arboviruses (dengue fever, Zika, chikungunya and Ross River) malaria as well as the seroprevalence of SARS-CoV-2.

Repeated regularly, these surveys allow the ASS-NC to capitalize on population indicators, to compare them according to socio-demographic characteristics, to identify groups at risk, to provide changes in health behaviors and to strengthen analytical capacities in order to adapt the guidelines for public policies and prevention programs.

DETAILED DESCRIPTION:
The "Barometre Santé Adulte" is an observational, descriptive and cross-sectional study whose data collection will take place in New Caledonia.

For this study the sampling is based on the 2019 population census, according to a 3-stage stratified sample design. In total, the main sample will consist of approximately 5,500 people (first phase) and the sub-sample will consist of 1,800 people (second phase).

The participation rate is estimated at 60%. Data collection will take place from February to May at the people's place drawn according to two steps:

* Firstly, investigators will carry out a questionnaire with the people who gave their informed consent as well as taking physical measurements: height, weight, abdominal circumference and blood pressure. In addition to the socio-demographic characteristics of the respondents, the questionnaire deals with several health topics: consumption of psychoactive substances, diet, physical activity, health status and access to care, screening, oral health, driving motor vehicle risk, sexual health, mental health, etc. The time taken to complete the questionnaire is estimated at one hour.
* Secondly, and for a sub-sample of 1,800 people, nurses will come back to the people's places who volunteer to take a venous blood test: blood sugar, total cholesterol, HbA1c, serum creatinine, CBC and serology of diseases transmitted by mosquitoes (dengue, chikungunya, Zika and Ross River, malaria).

All the data collected will be entered on a tablet in the eSTEPS application. The analysis of data (R Studio software) and the drafting of the report will be carried out by ASSNC staff. The first results are expected for the second half of 2022.

ELIGIBILITY:
Inclusion Criteria:

* Individuals informed of the conduct of the research and having given their written consent to participate in the study (questionnaire and taking physical measurements);
* Individuals between the ages of 18 and 64;
* Individuals residing in New Caledonia in so-called "ordinary" housing under their main residence at the last population census in 2019;

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Tourists and transients staying in New Caledonia for less than 6 months at the time of the investigation;
* People who are not intellectually fit to answer the questionnaire;
* Persons subject to guardianship, curatorship or any other legal incapacity;
* For the second phase of the study will be excluded people describing a febrile syndrome;

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5471 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
To know the prevalence of the main risk factors chronic diseases (obesity, diabetes, high blood pressure, high cholesterol and kidney failure) in the adult population of New Caledonia aged 18 to 64 using the WHO STEPS survey method. | Within a year after recruiting the participant
  In order to measure the prevalence of the main risk factors chronic diseases, WHO STEPS method will be used. This questionnaire is a 3 steps method, the first steps is a questionnaire mainly based on medical history and health behaviors. The second steps is associated with taking physical measurements such as weight, height, blood pressure, waist size. The last steps concerned only the experimental group "the sub-sample" for which some blood sample will be drawn out for the detection of elevated levels of blood glucose, HbA1c, total cholesterol and serum creatinine.

SECONDARY OUTCOMES:
Health behaviors of the target population using the first step of the WHO STEPS survey method. | Within a year after recruiting the participant
  To correlate health data and everyday behaviors of the target population in order to show a trend in causal effect, in order to have specific health indicators up to date
To calculate the cardiovascular risk of the New Caledonian population using the SCORE projet | Within a year after recruiting the participant
  To calculate the cardiovascular risk based on systolic blood pressure, sex, smoking status and cholesterol level.
Seroprevalence of infectious diseases | Within a year after recruiting the participant
  To Determine the seroprevalence of dengue, Zika, chikungunya and Ross River arboviruses in New Caledonia, the seroprevalence against the malaria agent as well as the seroprevalence of SARS-CoV-2.

CONTACTS AND LOCATIONS:
Locations (1):
- Agence Sanitaire et Sociale Nouvelle Calédonie, Noumea, New Caledonia

IPD SHARING:
Plan to Share IPD: Yes
Data will be share in new caledonia open data website. Data will be cleaned and anonymized prior sharing in on the open data
Supporting Information: SAP
Time Frame: within 1 year after the study end
Access Criteria: Open access
URL: http://data.gouv.nc/pages/accueil/?flg=fr